CLINICAL TRIAL: NCT03659786
Title: Cumulus Cell Messenger Ribonucleic Acid (mRNA) Analysis as Oocyte Quality Marker in the Fertility Lab in a Prospective Single-center Study
Brief Title: Single-center Prospective Cumulus Cell Test Study
Acronym: CC-Test
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BUN143201318000
Record Dates: First submitted 2018-09-03; First posted 2018-09-06 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Pregnancy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CC-Test diagnosis and Day 3 transfer (Experimental): Patients undergo the standard ART treatment, as prescribed by the treating physician, with standard morphology based scoring of the embryos + the extra cumulus cell based diagnosis and transfer of the best embryo based on morphology and CC diagnosis on day 3 of embryo growth (cleavage stage embryo)
  Interventions: Other: CC-Test
- Day 3 transfer control group (No Intervention): Patients undergo the standard ART treatment, as prescribed by the treating physician, with standard morphology based scoring of the embryos and transfer of the best embryo based on day 3 of embryo growth (cleavage stage embryo)
- Day 5 transfer control group (No Intervention): Patients undergo the standard ART treatment, as prescribed by the treating physician, with standard morphology based scoring of the embryos and transfer of the best embryo based on day 5 of embryo growth (blastocyst stage embryo)

INTERVENTIONS:
Other: CC-Test — Classification of the oocyte/embryo based on the expression pattern observed in the cumulus cells
  Arms: CC-Test diagnosis and Day 3 transfer

SUMMARY:
Performing an additional non-invasive oocyte diagnostic test based on cumulus cell gene expression could improve the outcome of the ART cycle

ELIGIBILITY:
Inclusion Criteria:

* scheduled for intracytoplasmatic sperm injection (ICSI) and single or double embryo transfer on day 3
* patients down regulated with gonadotropin-releasing hormone (GnRH) antagonist and stimulated with Highly Purified human Menopausal Gonadotropin (HP-hMG)
* undergoing first or second IVF or ICSI cycle with transfer
* Body Mass Index (BMI) between 17 and 33.
* regular menstrual cycle (between 24 and 35 days)

Exclusion Criteria:

* smokers (> 10 cigarettes per day)
* patients requesting Pre-implantation Genetic Diagnosis (PGD)
* patients with polycystic ovary syndrome (PCOS), or severe endometriosis (AFS stage 3-4)
* couples where the partner has an extremely low sperm count e.g.: extreme oligo-astheno-teratozoospermia (OAT) (< 100.000/ml) or scheduled for testicular sperm extraction (TESE)
* results of eventual preceding cycles may not indicate a known genetic disease, or low ovarian response or an oocyte maturation defect

Max Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-10 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy as observed by ultrasound | 2 months after embryo transfer
  This observation is routinely performed by the treating physician for every patient undergoing standard ART treatment and is thus available from the fertility center database

SECONDARY OUTCOMES:
Positive beta-hCG Pregnancy as observed by serum analysis | 12-17 days after embryo transfer
  This observation is routinely performed by the treating physician for every patient undergoing standard ART treatment and is thus available from the fertility center database
Live birth by questionnaire | at least 9 months after embryo transfer
  This observation is routinely performed by the study nurses of the fertility center for every patient undergoing standard ART treatment and is thus available from the fertility center database.This measurement does not include a scale, there is either a child born or not. The date of delivery and the gender of the child are asked together with eventual complications.
Cumulative pregnancy | 2 years after embryo transfer
  This is the compilation of the data gathered in outcome 1 and 3 for eventual consecutive cycles. This observation is routinely performed by the study nurses of the fertility center for every patient undergoing standard ART treatment and is thus available from the fertility center database.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Smitz, Prof. Dr., Study Director — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van Vaerenbergh I, Adriaenssens T, Coucke W, Van Landuyt L, Verheyen G, De Brucker M, Camus M, Platteau P, De Vos M, Van Hecke E, Rosenthal A, Smitz J. Improved clinical outcomes after non-invasive oocyte selection and Day 3 eSET in ICSI patients. Reprod Biol Endocrinol. 2021 Feb 19;19(1):26. doi: 10.1186/s12958-021-00704-5. PMID 33608027